CLINICAL TRIAL: NCT00611689
Title: A Phase I Study to Determine the Safety of Imatinib in Combination With PTK787/ZK222584 in Patients With Refractory and/or Advanced Solid Tumors
Brief Title: Imatinib and PTK787/ZK222584 in Refractory and/or Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 51
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Refractory Malignancy; Solid Tumors
Keywords: Refractory Malignancy; Solid Tumors; PTK787; ZK222584
MeSH Terms: conditions — Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Imatinib and PTK/ZK222584
  Interventions: Drug: Imatinib and PTK/ZK222584

INTERVENTIONS:
Drug: Imatinib and PTK/ZK222584 — Imatinib and PTK/ZK will each be administered orally daily. Two dose levels of imatinib (400 mg and 600 mg) will be tested with 4 dose levels of PTK/ZK (250 mg, 500 mg, 750 mg, and 1000 mg). 3 patients will be accrued at each individual dose level. If dose-limiting toxicities are reported in ≤ 1/3 patients, the dose level will be expanded to 6 patients. If dose-limiting toxicities are reported in < 2/6 patients, then dose escalation will continue. If ≥ 2/6 patients experience dose-limiting toxicity, the next lower dose will be considered the maximum tolerated dose and will be expanded to a total of 12 patients. There will be no intrapatient dose escalations. Patients may continue to receive treatment until unacceptable toxicity or disease progression is encountered.

SUMMARY:
In this phase I study, the investigators will determine the maximum tolerated doses of imatinib and PTK/ZK administered in two different dose schedules. Due to the different mechanisms of action and the minimally-overlapping toxicity profiles of these two novel oral agents, it is hoped that a combination regimen incorporating both compounds will produce increased activity without enhanced toxicity. After completion of this phase I study, the investigators propose a follow-up phase II study in patients with previously treated metastatic renal cell cancer - where VEGF and PDGF appear to play important roles in the malignant phenotype - to determine the antitumor efficacy of the recommended dose of this combination regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy-proven, advanced, incurable solid tumors refractory to standard treatment or for which there is no known standard treatment.
2. ECOG performance status 0 or 1.
3. Life expectancy of at least three months.
4. At least three weeks from any previous chemotherapy or 4 weeks from all investigational treatment
5. Completed any previous radiotherapy at least two weeks prior to study entry.
6. Adequate end organ function, defined as the following: total bilirubin < 1.5 x ULN, creatinine < 1.5 x ULN, ANC > 1500/µL, platelets > 100,000/µL.
7. Serum bilirubin <= 1.5 x the institutional upper-limit of normal and alkaline phosphatase, AST (SGOT), and ALT (SGPT) <= 2.5 x the institutional upper-limit of normal (within 7 days prior to initial treatment).
8. Hemoglobin >= 9 gm/dL (may be transfused or receive erythropoietin to maintain or exceed this level).
9. Patients with a history of brain metastases are eligible, but only if they have had previous treatment for the metastases and these are inactive and asymptomatic at the time of enrollment in this study.
10. Patients must be able to understand the nature of this study and give written informed consent.
11. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug. Oral, injectable, and injection contraceptives should not be considered effective as they may be affected by cytochrome P450 interactions.
12. Must have evaluable-disease
13. Must be > 18 years of age.
14. Patients may have received prior systemic chemotherapy, i.e. there is no limit on the number of prior regimens the patient may have received.

Exclusion Criteria:

1. Female patients who are pregnant or are lactating.
2. History of acute myocardial infarction within 6 months. In addition, patients are ineligible if they have clinically significant cardiovascular disease (e.g. uncontrolled hypertension, unstable angina), New York Heart Association grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or > grade II peripheral vascular disease.
3. Patients with a prior malignancy (except for adequately treated basal-cell or squamous-cell skin cancers, in situ carcinomas, or low grade [Gleason score 3+3 or less] localized prostate cancer) in the past 5 years will be excluded.
4. Patients with active concurrent infections or patients with serious underlying medical conditions will be excluded from the study.
5. Women who are pregnant or lactating are ineligible. All men and women of reproductive potential must agree to use effective contraception while receiving treatment in this study. (See 3.1.11)
6. Patients who are concurrently using phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, systemic retinoids, or St. John's Wort are ineligible.
7. Patients who have had a prior grade 4 thromboembolic event are ineligible. Patients who have had a grade 3 thromboembolic event are ineligible unless they have an in-range INR (usually between 2 and 3) on a stable dose of low molecular weight heparin or unfractionated heparin. In addition, patients who have clinical or radiologic evidence of clots in the renal veins, inferior vena cava, hepatic veins, or portal vein are ineligible. Since warfarin is metabolized through the CYP450 system, no therapeutic anticoagulation with warfarin (e.g. Coumadin or Coumadine) will be permitted in patients participating in this study. As an alternative, therapeutic anticoagulation may be accomplished using low-molecular weight heparin (e.g. Lovenox) or heparin. Mini-Dose Coumadin (e.g. 1 mg qd) is permitted for prophylaxis of central venous catheter thrombosis, at the discretion of the treating physician. In general, the use of Coumadin is discouraged on this protocol.
8. Major surgical procedure, open biopsy; or significant traumatic injury within 28 days or anticipation of need for major surgical procedure during the course of the study.
9. Patients with PEG or G-tubes are ineligible.
10. Proteinuria; if > 1+ on dipstick at baseline patients must have 24-hour urine collection. Patients with > 500mg protein/24 hrs are ineligible. (See Appendix A - Evaluation and Management of Proteinuria).
11. Any nonhealing wound, ulcer, or bone fracture.
12. Any clinical evidence or history of a bleeding diathesis or coagulopathy.
13. Participation in another experimental drug study within 28 days of starting treatment.
14. History of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications.
15. Presence of poorly controlled hypertension (as defined by the treating clinician) If a patient's condition is deteriorating, laboratory evaluations should be repeated < 48 hours prior to initiation of therapy.
16. Prior VEGF therapy.
17. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK787/ZK 222584 (i.e. ulcerative disease, uncontrolled nausea, vomiting diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-07; Primary Completion 2008-01 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
MTD and the recommended phase II doses of imatinib and PTK/ZK administered daily every 28 days | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States